CLINICAL TRIAL: NCT00366535
Title: Neurotropin Treatment of Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health Clinical Center (CC) (NIH); University of Michigan (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 060229; NCT00366535 (Registry Identifier: ClinicalTrials.gov); 06-NR-0229 (Other: NIH)
Record Dates: First submitted 2006-08-18; First posted 2006-08-21 (Estimated); Results first posted 2018-06-04 (Actual); Last update posted 2018-06-27 (Actual); Status verified 2018-05

CONDITIONS: Fibromyalgia
Keywords: Muscle Pain; Fibrositis Allodynia; Stiffness; Tender Points; Fibromyalgia
MeSH Terms: conditions — Fibromyalgia; Myalgia | interventions — neurotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (2):
- Placebo first, then Neurotropin (G-1) (Active Comparator): Double blind cross-over study: receive Placebo for 12 weeks and then Neurotropin for 12 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others blind.
  Interventions: Drug: Placebo; Drug: Neurotropin
- Neurotropin first, then Placebo (G-2) (Active Comparator): Double blind cross-over study: receive Neurotropin for 12 weeks and then Placebo for 12 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others
  Interventions: Drug: Placebo; Drug: Neurotropin

INTERVENTIONS:
Drug: Placebo — 4 tabs b.i.d.
  Other Names: Drug A
Drug: Neurotropin — 4 tabs b.i.d.
  Other Names: Drug B

SUMMARY:
This study will examine the safety and effectiveness of the experimental drug, neurotropin, for preventing or easing pain associated with fibromyalgia. A disorder that primarily affects women, fibromyalgia causes widespread aching and stiffness in muscles. Neurotropin has been used in Japan for many years to treat various chronic painful conditions, including fibromyalgia.

Women with fibromyalgia who have been treated unsuccessfully with standard therapy may be eligible for this study. Patients must have a history of widespread pain for more than half of the days in each of the three months before they enter the study. Candidates are screened with a medical history, physical examination, blood and urine tests, questionnaires and an electrocardiogram (EKG).

Participants take their usual medications for fibromyalgia in addition to either neurotropin or a placebo (look-alike medicine with no active ingredient). At 6 weeks and 12 weeks into the study, they return to the NIH Clinical Center for evaluation of their sensitivity to pain and level of physical capability. After 12 weeks, study subjects "cross-over" their medication; that is, patients who took neurotropin for the first 12 weeks of the study take placebo for the next 12 weeks, and vice-versa. Again, after 6 and 12 weeks, patients return for evaluation.

Participants have blood and urine tests six times during the study and complete questionnaires each week about their pain, symptoms, and activities.

DETAILED DESCRIPTION:
Fibromyalgia is a relatively common disorder, which occurs predominantly in women, that is characterized by widespread aching and stiffness in muscles. Although there have been numerous studies of fibromyalgia, its etiology has remained unclear, but it is generally believed that central pain processing abnormalities are involved. Neurotropin, a non-protein extract of inflamed cutaneous tissue from rabbits inoculated with vaccinia virus, has been used extensively in Japan for many years to treat a variety of chronic painful conditions, including fibromyalgia. This present protocol is a double blind, placebo-controlled, crossover study designed to examine the clinical efficacy of Neurotropin in treating women (neither pregnant nor lactating) suffering from fibromyalgia without evidence of any other cause of their complaint of pain. Patients must meet the American College of Rheumatology (ACR) diagnostic criteria for fibromyalgia and must agree to maintain a stable therapeutic regimen throughout the 25-week study.

ELIGIBILITY:
INCLUSION CRITERIA:

Subjects will be drawn from a cohort of well-characterized female fibromyalgia patients who were under the care of Dr. Daniel. J. Clauw when he was at Georgetown University. All patients must continue to meet the criteria established by the ACR for diagnosis of fibromyalgia, and must have been treated unsuccessfully with a current standard therapeutic regimen. The criteria are (A) a history of widespread pain (in all quadrants and back) for more than half of the days in each of the prior three months and (B) the required number,11, of tender points of 18 test sites (indicated in Figure 1), which will be determined during the initial physical examination (see below). They must give informed consent to participate in this study. It is anticipated that almost all patients will be residents of Washington, D.C. area and that they will be able to travel to NIH for necessary preliminary studies and subsequent required evaluations. To be admitted to this study, patients must be willing to continue using only their present medications (including antidepressants) or other forms of care related to the control of fibromyalgia symptoms during the course of the study. The average score on the FIQ for patients seen in tertiary care settings is about 50 (with 100 being the maximum, a higher score indicating a greater impairment of health) and we will include only those patients in whom the FIQ score is greater than 30 at the initial evaluation.

EXCLUSION CRITERIA:

Pregnant and lactating women are excluded because of the bodily changes that would occur during the study. As indicated above, a pregnancy test will be performed in women of childbearing age (up to age 55). The combination of widespread musculoskeletal pain, high tender point count, and non-restorative sleep are usually sufficient criteria for the diagnosis of fibromyalgia and the patients referred for this study will have been well characterized in the Fibromyalgia Clinic at Georgetown University or by the referring physician. We will, however, by history, physical examination, screening laboratory studies and examination of the patient s medical records confirm the absence of any evidence for peripheral neuropathies, entrapment syndromes, neurologic disorders or metabolic/endocrine disorders, such as untreated hypothyroidism, as well as the rheumatoid disorders that might be confused with fibromyalgia and confound the study. Patients who have abnormal screening test results or who have traumatic or non-traumatic disorders to which pain may be attributed. Also, patients who have a positive HIV result will be excluded. Subjects with obviously impaired mental capacity that precludes informed consent and ability to provide adequate self-ratings are to be excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2006-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leorey N Saligan, C.R.N.P., Principal Investigator — National Institute of Nursing Research (NINR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dworkin RH, Fields HL. Fibromyalgia from the perspective of neuropathic pain. J Rheumatol Suppl. 2005 Aug;75:1-5. No abstract available. PMID 16078355
- [Background] Rowbotham MC. Is fibromyalgia a neuropathic pain syndrome? J Rheumatol Suppl. 2005 Aug;75:38-40. PMID 16078359
- [Background] Crofford LJ. The relationship of fibromyalgia to neuropathic pain syndromes. J Rheumatol Suppl. 2005 Aug;75:41-5. PMID 16078360
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-NR-0229.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Most patients were recruited by direct physician referral or through the Patient Recruitment and Public Liaison (PRPL) office. Potential subjects were screened for study eligibility at the NIH Clinical Center.
Pre-assignment Details: Patients with abnormal screening laboratory tests or had positive HIV test were excluded from study participation. Women who had positive urine pregnancy test were also excluded. Also patients with traumatic or non-traumatic pain disorders or had neurocognitive impairment making it challenging to obtain informed consent, were also excluded.
Groups:
- Study Drug A Then Study Drug B (G-1): Double blind cross-over study: received Placebo (4 tabs, b.i.d.) for 12 weeks and then Neurotropin (4 tabs, b.i.d.) for 12 weeks (after at least 1 week washout period). Assignment to each group was randomized by the NIH Clinical Center pharmacy. Study team and participants were all blinded.
- Study Drug B First, Then Study Drug A (G-2): Double blind cross-over study: received Study drug B (4 tabs, b.i.d.) for 12 weeks and then Study drug A (4 tabs, b.i.d.) for 12 weeks (after at least 1 week washout period). Assignment to each group was randomized by the NIH CC pharmacy. Study team and participants were blinded.
Period: First Phase: 12 Weeks
Arm/Group | Study Drug A Then Study Drug B (G-1) | Study Drug B First, Then Study Drug A (G-2)
Started | 27 | 29
Completed | 24 | 21
Not Completed | 3 | 8
Not completed — Adverse Event | 1 | 3
Not completed — Withdrawal by Subject | 2 | 5
Period: Washout Period (at Least a Week)
Arm/Group | Study Drug A Then Study Drug B (G-1) | Study Drug B First, Then Study Drug A (G-2)
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0
Period: Second Phase: 12 Weeks
Arm/Group | Study Drug A Then Study Drug B (G-1) | Study Drug B First, Then Study Drug A (G-2)
Started | 24 | 21
Completed | 21 | 18
Not Completed | 3 | 3
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo First, Then Neurotropin (G-1): Double blind cross-over study: receive Placebo (4 tabs, b.i.d.) for 12 weeks and then Neurotropin (4 tabs, b.i.d.) for 12 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others blind.
- Neurotropin First, Then Placebo (G-2): Double blind cross-over study: receive Neurotropin (4 tabs, b.i.d.) for 12 weeks and then Placebo (4 tabs, b.i.d.) for 12 weeks (after at least 1 week washout period). Assignment to each group was in random order, selected by the pharmacy with all others blind.
- Total: Total of all reporting groups
Arm/Group | Placebo First, Then Neurotropin (G-1) | Neurotropin First, Then Placebo (G-2) | Total
Number analyzed (Participants) | 29 | 27 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (12.6) | 41.7 (12.9) | 44.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Because fibromyalgia is much more common in women and because there are significant gender differences in the clinical characteristics of the disorder, only women will be included in the study.
  Participants
    Female | 29 | 27 | 56
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 27 | 20 | 47
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29 | 27 | 56

OUTCOME MEASURES:

1. Primary Outcome: Fibromyalgia Impact Questionnaire
Description: The Fibromyalgia Impact Questionnaire (FIQ) is a brief 10-item self-administered measure to assess 3 areas of fibromyalgia (FM): function, overall impact, and symptoms. The total FIQ score was the primary outcome of the study. The total FIQ score is the sum of the 3 areas measured in the FIQ. The maximum possible total FIQ score is 100, with a minimum score of 10. The average FM patient scores about 50, severely afflicted FM patients are usually 70 and above. Data analysis is ongoing from data collected from study completers.
Time Frame: 25 weeks
Population: Total 56 patients enrolled, and 39 patients completed the study. 17 patients withdrawn from the study. Three of 39 patients were excluded from the data analysis because there had missing FIQ scores at Baseline and/or Week 12. The data from the study of the 36 participants with complete data sets was analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- FIQ Before Placebo Treatment First in G-1; FIQ Before Placebo Treatment Second in G-2: FIQ of this group was determined before the 12 week-treatment with Placebo.
- FIQ After Placebo Treatment First in G-1: This group received Placebo 4 tabs b.i.d. for 12 weeks first. FIQ was determined at the end of the 12 week-treatment with Placebo.
- FIQ Before Neurotropin Treatment Second in G-1; FIQ Before Neurotropin Treatment First in G-2: FIQ of this group was determined before the 12 week-treatment with Neurotropin.
- FIQ After Neurotropin Treatment Second in G-1: This group received Neurotropin 4 tabs b.i.d. for 12 weeks after at least 1 week "washout" period following the first 12 week interval on placebo. FIQ was determined at the end of the 12 week-treatment with Neurotropin.
- FIQ After Neurotropin Treatment First in G-2: This group received Neurotropin 4 tabs b.i.d. for 12 weeks first. FIQ was determined at the end of the 12 week-treatment with Placebo.
- FIQ After Placebo Treatment Second in G-2: This group received Placebo 4 tabs b.i.d. for 12 weeks after at least 1 week "washout" period following the first 12 week interval on placebo. FIQ was determined at the end of the 12 week-treatment with Placebo.
Arm/Group | FIQ Before Placebo Treatment First in G-1 | FIQ After Placebo Treatment First in G-1 | FIQ Before Neurotropin Treatment Second in G-1 | FIQ After Neurotropin Treatment Second in G-1 | FIQ Before Neurotropin Treatment First in G-2 | FIQ After Neurotropin Treatment First in G-2 | FIQ Before Placebo Treatment Second in G-2 | FIQ After Placebo Treatment Second in G-2
Number analyzed (Participants) | 20 | 20 | 20 | 20 | 16 | 16 | 16 | 16
units on a scale | 49.9 (1.8) | 37.5 (3.7) | 39.9 (3.4) | 33.4 (4.1) | 47.7 (2.1) | 28.8 (4.5) | 30.1 (4.1) | 32.8 (3.6)

ADVERSE EVENTS:
Time Frame: The adverse event data was collected during the study period for 6 to 7 months.
Groups:
- Placebo Treatment First in G-1: This group received Placebo 4 tabs b.i.d. for the first 12 weeks.
- Neurotropin Treatment Second in G-1: This group received Neurotropin 4 tabs b.i.d. for 12 weeks after at least 1 week "washout" period following the first 12 week interval on Placebo.
- Neurotropin Treatment First in G-2: This group received Neurotropin 4 tabs b.i.d. for the first 12 weeks.
- Placebo Treatment Second in G-2: This group received Placebo 4 tabs b.i.d. for 12 weeks after at least 1 week "washout" period following the first 12 week interval on Neurotropin.
Arm/Group | Placebo Treatment First in G-1 | Neurotropin Treatment Second in G-1 | Neurotropin Treatment First in G-2 | Placebo Treatment Second in G-2
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/29 | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/29 | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 3/56 | 1/29 | 3/27 | 1/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Treatment First in G-1 (N=56) | Neurotropin Treatment Second in G-1 (N=29) | Neurotropin Treatment First in G-2 (N=27) | Placebo Treatment Second in G-2 (N=27)
Abnormality of liver function test (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Increased in plasma levels of ALT, AST and LDH, and creatinine kinase
Chest pain and Abnormal HB (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) — Chest pain followed by dizziness, shortness of breath and weakness, abnormal heart beat
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) — Increased of pain
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Caused dizziness, headache and difficulty walking

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes